CLINICAL TRIAL: NCT01109589
Title: Respiratory Tract Infections and Prescription Drugs in Children and in Pregnancy - a Study From Norwegian General Practice
Brief Title: Respiratory Tract Infections and Prescription Drugs in Children and in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Responsible Party: Professor Morten Lindbæk, MD, PhD, Antibiotic Centre for Primary Care, University of Oslo
Other Study IDs: ASP-UIO-2010
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Respiratory Tract Diagnoses (ICPC-2); Prescriptions of Antibiotics by General Practitioners; Prescriptions of ATC J01 and R Drugs in Participants
Keywords: antibiotics; prescriptions; pregnancy; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children aged 0-2 yrs
- Women aged 15-60 yrs

SUMMARY:
The main objective is to investigate the incidence of Respiratory Tract Infections (RTIs) and antibiotic prescriptions in children and during pregnancy, the different drugs chosen by their doctors according to diagnosis, and compliance by patients. Further to investigate the possible effect of antibiotic use during pregnancy on RTIs and antibiotics and respiratory drug prescriptions in children the first two years after birth.

Specific study objectives:

* RTIs and antibiotic prescriptions in pre-school children

  * Frequency of diagnoses and antibiotic prescriptions
  * The proportion of broad spectrum antibiotics chosen
* Prescription patterns and treatment compliance during pregnancy

  * Incidence of diagnoses, compared with not pregnant patients
  * Choice of antibiotics in RTIs
  * Prescription collection from pharmacies
* Antibiotics and respiratory medication in children aged 0-2 yrs

  * Compare prevalence in children of mothers with frequent RTIs/antibiotic prescriptions during pregnancy and prevalence in children of mothers with few or no consultations during pregnancy
  * Incidence of wheezing and asthma diagnoses and incidence og respiratory prescription drugs when the mother has received antibiotics in pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Contact with general practitioner in the time of registration

Exclusion Criteria:

* Men (except children aged 0-2 yrs)
* Women in ages 2-14 and above 60 yrs

Max Age: 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Contacts with general practitioner in different parts of Norway. Women aged 15-60 yrs and children 0-2 yrs are selected.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2004-12; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antibiotic Centre for Primary Care, University of Oslo, Oslo, Norway